CLINICAL TRIAL: NCT03831750
Title: Assessing the Effectiveness of a Stress Reduction Intervention in Inflammatory Bowel Disease (IBD): a Prospective Randomized Controlled Trial (RCT)
Brief Title: Assessing the Effectiveness of a Stress Reduction Intervention in Inflammatory Bowel Disease (IBD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00082125; Pro00079377
Record Dates: First submitted 2019-02-04; First posted 2019-02-06 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Inflammatory Bowel Diseases; Remission; Perceived Stress
Keywords: ulcerative colitis; remission; perceived stress; fecal calprotectin; salivary stress biomarker; psychological stress; stress reduction; Crohn's disease; Inflammatory bowel diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Stress, Psychological; Crohn Disease

STUDY DESIGN:
Who Masked: Participant
Masking Description: Sealed envelopes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stress Reduction Intervention (Experimental): Participants will receive the standard of care for IBD and training and access to an online stress reduction intervention.
  Interventions: Other: Stress Reduction Intervention
- Control (No Intervention): Participants will receive the standard of care for IBD.

INTERVENTIONS:
Other: Stress Reduction Intervention — The tri-component intervention is comprised of guided videos for breath-work (5-15 min), stretching (5-15 min), and meditation (10-30 min). The intervention will be delivered online via an access restricted website.
  Arms: Stress Reduction Intervention

SUMMARY:
The investigators have designed a guided, online, tri-component, stress reduction intervention for participants with inflammatory bowel diseases.

DETAILED DESCRIPTION:
In a randomized controlled trial, the investigators assessed the impact of an online, 3-month stress reduction intervention (yoga, breathwork, and meditation). The primary outcome was the change in Cohen's Perceived Stress Scale (PSS) between the control and intervention arms. The following secondary outcomes were also assessed: anxiety, depression, IBD disease activity (e.g., changes in CRP, fecal calprotectin, medication, hospitalization, or surgery), serum inflammatory markers, serum and salivary markers of stress, stress-resilience, and health- related quality of life. Participant satisfaction and adherence to the intervention were also evaluated.

ELIGIBILITY:
Inclusion Criteria (RCT):

* Adults (≥18 years)
* with IBD in remission (UC - partial Mayo <2 and fecal calprotectin <250 μg/g; CD regular HBI <5 or CRP <8)
* on stable therapy for the past 3 months
* the last flare <24 months prior to enrollment
* PSS-10 score ≥ 7 at time of screening

Inclusion Criteria (Substudy):

* Adults (≥18 years)
* IBD
* on stable therapy for the past 3 months.

Exclusion Criteria (RCT or Substudy):

* Major medical co-morbidity
* Steroid use in past 3 months
* Clostridium difficile infection in the last 3 months
* Unstable dose of psychiatric medications for the last 3 months
* Inability to provide informed written consent
* Severe psychiatric disorders (HADS scores >10 or suicidal ideation)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2019-02-22 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Perceived stress | 3 months
  Between group changes in the stress index from baseline to end of study using the Cohen's Perceived Stress Scale (PSS)-10 item. Summed scores range from 0-40 where lower scores are associated with less perceived stress compared to higher scores.

SECONDARY OUTCOMES:
Mental health | 3 months
  Change from baseline to end of study using the Hospital and Anxiety Depression Scale (HADS). Summed scores (range: 0-21) are separate for anxiety and depression; lower scores are assocated with less perceived anxiety or depression.
Health-related quality of life | 3 months
  Change from baseline to end of study using the: (1) Short IBD Quality of Life Questionnaire (SIBDQ). Scores (range 1-7) for the 7 questions are summed where higher scores related to a higher perceived health-related quality of life.
Markers of inflammation and stress | 3 months
  Changes from baseline to end of study for 6 serum pro- and anti-inflammatory immune biomarkers relevant to IBD (IL-10, IL-12, IL-1ß, IL-4, IL-6, TNF-α) and markers of stress, including CABS1 and cortisol, with the Connor Davidson Resilience Scale (score range: 0 to 100). Higher scores with the Connor Davidson Resilience Scare are indicative of greater stress resiliency.
IBD levels of activity | 3 months
  Changes from baseline to end of study for fecal calprotectin and Partial Mayo Score (score range 0-9; lower scores mean less or no disease activity) or the Harvey Bradshaw Index (HBI) (range=0-16+; where lower scores indicate less or no disease activity).

CONTACTS AND LOCATIONS:
Overall Officials: Farhad Peerani, MD, Principal Investigator — University of Alberta; Puneeta Tandon, MD, MSc, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Ritz T, Rosenfield D, St Laurent CD, Trueba AF, Werchan CA, Vogel PD, Auchus RJ, Reyes-Serratos E, Befus AD. A novel biomarker associated with distress in humans: calcium-binding protein, spermatid-specific 1 (CABS1). Am J Physiol Regul Integr Comp Physiol. 2017 Jun 1;312(6):R1004-R1016. doi: 10.1152/ajpregu.00393.2016. Epub 2017 Apr 5. PMID 28381457
- [Background] Bernstein CN, Singh S, Graff LA, Walker JR, Miller N, Cheang M. A prospective population-based study of triggers of symptomatic flares in IBD. Am J Gastroenterol. 2010 Sep;105(9):1994-2002. doi: 10.1038/ajg.2010.140. Epub 2010 Apr 6. PMID 20372115
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391
- [Derived] Peerani F, Watt M, Ismond KP, Whitlock R, Ambrosio L, Hotte N, Mitchell N, Bailey RJ, Kroeker K, Dieleman LA, Siffledeen J, Lim A, Wong K, Halloran BP, Baumgart DC, Taylor L, Raman M, Madsen KL, Tandon P. A randomized controlled trial of a multicomponent online stress reduction intervention in inflammatory bowel disease. Therap Adv Gastroenterol. 2022 Sep 27;15:17562848221127238. doi: 10.1177/17562848221127238. eCollection 2022. PMID 36187365